CLINICAL TRIAL: NCT03661983
Title: A Randomized, Placebo-controlled Trial to Evaluate the Long-term (ie, Maintenance) Efficacy of Oral Aripiprazole in the Treatment of Pediatric Subjects With Tourette's Disorder
Brief Title: Trial to Evaluate the Long-term Efficacy of Oral Aripiprazole in the Treatment of Pediatric Participants With Tourette's Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of feasibility for completion of the trial within a reasonable time frame.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-14-204; 2018-002270-48 (EudraCT Number)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Tourette's Disorder (TD)
Keywords: Aripiprazole; Tourette's Disorder; Pediatric
MeSH Terms: conditions — Tourette Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Open Label Stabilization Phase: Aripiprazole (Experimental): Participants began treatment with aripiprazole at a 2.0 mg/day dose, with the dose titrated to 5.0 mg/day after 2 days. Subsequent dose adjustments were based on the participant's weight to achieve optimum control of tics up to the maximum recommended doses based on the United States Labeling, up to Week 8 and then continued on the most stabilized dose up to minimum Week 14 or maximum Week 20. Participants who met stabilization criteria were randomized to Double-blind Randomization Phase.
  Interventions: Drug: Aripiprazole
- Double Blind Phase: Aripiprazole Full Dose (Experimental): Participants who met stabilization criteria and randomized to receive full dose of aripiprazole i.e. 5 mg or 10 mg for <50 kg participants,and 10 mg or 20 mg for >50 kg participants (2 tablets a day), based on stabilized dose in open-label stabilization phase, up to 12 weeks in Double-Blind Phase.
  Interventions: Drug: Aripiprazole
- Double Blind Phase: Aripiprazole Half Dose (Experimental): Participants who met stabilization criteria and randomized to receive half dose of aripiprazole i.e. 2 mg or 5 mg for <50 kg participants, and 5 mg or 10 mg for >50 kg participants (2 tablets a day), based on stabilized dose in open-label stabilization phase, up to 12 weeks in Double-Blind Phase.
  Interventions: Drug: Aripiprazole
- Double Blind Phase: Placebo (Placebo Comparator): Participants who met randomization criteria and randomized to receive aripiprazole matching-placebo tablets, 2 daily, orally, up to 12 weeks in Double-Blind Phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Participants received aripiprazole tablets, orally as per the regimen specified in the arm description.
  Other Names: OPC-14597
  Arms: Double Blind Phase: Aripiprazole Full Dose; Double Blind Phase: Aripiprazole Half Dose; Open Label Stabilization Phase: Aripiprazole
Drug: Placebo — Participants received aripiprazole matching-placebo tablets, orally as per the regimen specified in the arm description.
  Arms: Double Blind Phase: Placebo

SUMMARY:
To evaluate the long-term efficacy of oral aripiprazole in pediatric participants for the treatment of Tourette's Disorder (TD).

DETAILED DESCRIPTION:
This study will evaluate the long-term efficacy of oral aripiprazole in the treatment of pediatric participants with Tourette's Disorder (TD). The trial consists of 3 distinct phases: a pretreatment phase, open-label stabilization phase, and a double-blind randomized withdrawal phase.

ELIGIBILITY:
Inclusion Criteria:

* The participant is a male or female child or adolescent, 6 to 17 years of age (inclusive) at the time of signing the informed consent/assent.
* The participant meets current Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) diagnostic criteria for TD, documented at screening and made by an adequately trained clinician, as confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime Version.
* The participant has a Total Tic Score (TTS) ≥ 20 on the Yale Global Tic Severity Scale (YGTSS) at screening and baseline (Day 1).
* The participant, a caregiver, and the investigator must all agree that the presenting tic symptoms cause impairment in the participant's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships.
* Females of childbearing potential (all female participants ≥ 12 years of age and all female participants < 12 years of age if menstruation has started) must have a negative pregnancy test and must not be pregnant or lactating.
* Written informed consent must be obtained from the participant or a legally acceptable representative (eg, guardian or caregiver), in accordance with requirements of the trial site's institutional review board (IRB)/independent ethics committee (IEC) and local regulatory requirements, prior to the initiation of any protocol-required procedures. In addition, the participant, as required by the trial center's IRB/IEC, must provide informed assent at screening and as such must be able to understand that he or she can withdraw from the trial at any time.
* Ability, in the opinion of the principal investigator, of the participant and the participant's legally acceptable representative (e.g., guardian) or caregiver(s) to understand the nature of the trial and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, and discontinuation of prohibited concomitant medications, to read and understand the written word in order to complete participant-reported outcomes measures, and to be reliably rated on assessment scales.

Exclusion Criteria:

* The participant presents with a clinical presentation and/or history that is consistent with another neurologic condition that may have accompanying abnormal movements. These include, but are not limited to, the following: Transient tic disorder; Huntington's disease; Parkinson's disease; Sydenham's chorea; Wilson's disease; Mental retardation; Pervasive developmental disorder; Tardive dyskinesia; Traumatic brain injury; Stroke; Restless legs syndrome.
* The participant has a history of schizophrenia, bipolar disorder, or other psychotic disorder.
* Participants who receive psychostimulants for the treatment of attention-deficit hyperactivity disorder (ADHD) and who have developed and/or had exacerbations of the tic disorder after the initiation of stimulant treatment. (Note that participants with ADHD who are treated with psychostimulants and have not developed new tics or a worsening of their current tics can be included if all other enrollment obligations are met).
* The participant currently has a primary diagnosis that meets DSM-5 criteria for mood disorder.
* The participant has severe obsessive-compulsive disease, as evidenced by a Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) score > 16.
* The participant has taken aripiprazole within 1 month (30 days) of the screening visit.
* The participant has a history of neuroleptic malignant syndrome.
* Participant is a sexually active male or female of childbearing potential (FOCBP) (all female participants ≥ 12 years of age and all female participants < 12 years of age if menstruation has started) who will not agree to practice 2 acceptable methods of birth control or who will not remain abstinent during the trial and for 30 or 90 days following the last dose of Investigational medicinal product (IMP) for females and males, respectively. Abstinence will be permitted if it is confirmed and documented at every trial visit.
* The participant represents a significant risk of committing suicide based on history (suicide attempt in past 1 year).
* The participant has a body weight < 16 kg.
* Participants who have taken neuroleptic or antiparkinson drugs within 14 days prior to baseline.
* Participants requiring cognitive-behavioral therapy (CBT) for TD during the trial period. CBT for other nonexclusionary disorder must remain consistent through the trial.
* The participant has met DSM-5 criteria for any significant psychoactive substance use disorder within the past 3 months.
* A positive drug screen for cocaine, alcohol, or other drugs of abuse (excluding caffeine, nicotine, or prescribed psychostimulants for ADHD). Investigators can choose to repeat a positive drug screen one time during screening period after concurrence from the medical monitor. A second positive test for any drug of abuse would be exclusionary.
* Participant requiring medication not allowed per protocol.
* Use of any cytochrome P450 (CYP)2D6 and CYP3A4 inhibitors or CYP3A4 inducers within 14 days prior to baseline and for the duration of the trial.
* Other nutritional or dietary supplements and nonprescription herbal preparations for TD (eg, cannabinoids, N-acetylcysteine, omega-3 fatty acids, kava extracts, GABA supplements) within 7 days prior to baseline and for the duration of the trial, unless approved in advance by the medical monitor.
* The inability to swallow tablets or tolerate oral medication.
* Participant has participated in a clinical trial involving either study medication or interventional (non-medication) treatment for TD within the last 60 days.
* The following laboratory test results, vital signs and electrocardiogram (ECG) results are exclusionary: Platelets ≤ 75,000/mm^3; Hemoglobin ≤ 9 g/dL; Neutrophils, absolute ≤ 1000/mm^3; Aspartate aminotransferase > 3 × upper limit of normal (ULN) as defined by the central laboratory; Alanine aminotransferase > 3 × ULN as defined by the central laboratory; Creatinine ≥ 2 mg/dL; Diastolic blood pressure > 105 mmHg; Corrected QT interval ≥ 450 msec (males) or ≥ 470 msec (females) using the corrected QT interval for heart rate using Fridericia's formula

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, MS, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (42):
- United States (38):
  - Advanced Research Center, Anaheim, California
  - CT Trials - Riverside, Riverside, California
  - Syrentis Clinical Research, Santa Ana, California
  - Comprehensive Research Center, Norwich, Connecticut
  - Sarkis Clinical, Gainesville, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Eastern Research, Hialeah, Florida
  - Quest Pharmaceutical Services - Miami Research Associates, South Miami, Florida
  - Rothman Center for Pediatric Neuropsychiatry, St. Petersburg, Florida
  - Pediatric and Adolescent Neurodevelopment Associates, Atlanta, Georgia
  - Inova Clinical trials and Research Center, Fayetteville, Georgia
  - Baber Research Group, Naperville, Illinois
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Alivation, Lincoln, Nebraska
  - The NeuroCognitive Institute, Mount Arlington, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - Mood Disorders Consulting Medicine, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Quest Therapeutics of Avon Lake DBA Haidar Almhana Nieding, Avon Lake, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Charak Center for Health and Wellness, Garfield Heights, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - ClinMed Research Associates, Inc., Oklahoma City, Oklahoma
  - Rivus Wellness and Research Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - BioBehavioral Research of Austin, Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Psychiatric Medical Associates, Plano, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Aspen Clinical Research - Orem, Orem, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Clinical Research Partners - Richmond, Petersburg, Virginia
  - Core Clinical Research, Everett, Washington
  - Palouse Psychiatry & Behavioral Health, Spokane, Washington
- Canada (2):
  - Kids Clinic, Ajax, Ontario
  - Jodha Tishon Inc., Toronto, Ontario
- Hungary (2):
  - Vadaskert Alaptvany A Gyermekek Lelki Egeszsegeert, Budapest
  - Semmelweis Egyetem - I. sz. Gyermekgyógyászati Klinika, Budapest

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in Canada, the United States and Hungary from Oct 13, 2018 to Jun 30, 2020.
Pre-assignment Details: Pediatric participants with a diagnosis of Tourette's Disorder were enrolled in this to receive oral aripiprazole in an Open-label Stabilization Phase and a Double-blind Randomized Withdrawal Phase and then followed for safety up to 30 days post-last dose.
Period: Open Label Stabilization Phase
Arm/Group | Open Label Stabilization Phase: Aripiprazole | Double Blind Phase: Aripiprazole Full Dose | Double Blind Phase: Aripiprazole Half Dose | Double Blind Phase: Placebo
Started | 36 | 0 | 0 | 0
Completed | 25 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 2 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 3 | 0 | 0 | 0
Period: Double-blind Randomized Phase
Arm/Group | Open Label Stabilization Phase: Aripiprazole | Double Blind Phase: Aripiprazole Full Dose | Double Blind Phase: Aripiprazole Half Dose | Double Blind Phase: Placebo
Started | 0 | 9 | 8 | 8
Completed | 0 | 7 | 7 | 0
Not Completed | 0 | 2 | 1 | 8
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Disease Relapse | 0 | 0 | 0 | 6
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled Sample included all participants who entered the open-label stabilization phase.
Arm/Group | Open Label Stabilization Phase: Aripiprazole
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 32
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 9
  Hungary | 4
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse During the Double-blind Randomized Withdrawal Phase
Description: Relapse was defined as a loss of ≥ 50% of the improvement experienced during the open-label stabilization phase (i.e., improvement at the last assessment of Yale Global Tic Severity Scale (YGTSS) before randomization) on the Yale Global Tic Severity Scale Total Tic Score (YGTSS TTS). YGTSS provides an evaluation of the number, frequency, intensity, complexity, and interference of motor and phonic symptoms.
Time Frame: From Randomization up to 12 weeks in Double-blind Randomized Withdrawal Phase
Population: Intent to Treat (ITT) Sample included all participants who were randomized and received at least 1 dose of randomized investigational medicinal product (IMP) were included in this dataset and were analyzed according to the treatment group they were randomized to.
Measure: Number; unit: percentage of participants
Arm/Group | Double Blind Phase: Aripiprazole Full Dose | Double Blind Phase: Aripiprazole Half Dose | Double Blind Phase: Placebo
Number analyzed (Participants) | 9 | 8 | 8
percentage of participants | 0.0 | 0.0 | 75.0

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose of study drug (Up to approximately 36 weeks)
Description: Open-label Safety Sample included all participants that had administered at least 1 dose of IMP during the open-label stabilization phase.
  Randomized Safety Sample included all participants who received at least 1 dose of randomized IMP during the double-blind randomized withdrawal phase were included and analyzed according to the treatment received.
Arm/Group | Open Label Stabilization Phase: Aripiprazole | Double Blind Phase: Aripiprazole Full Dose | Double Blind Phase: Aripiprazole Half Dose | Double Blind Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 17/36 | 3/9 | 3/8 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Stabilization Phase: Aripiprazole (N=36) | Double Blind Phase: Aripiprazole Full Dose (N=9) | Double Blind Phase: Aripiprazole Half Dose (N=8) | Double Blind Phase: Placebo (N=8)
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Stabilization Phase: Aripiprazole (N=36) | Double Blind Phase: Aripiprazole Full Dose (N=9) | Double Blind Phase: Aripiprazole Half Dose (N=8) | Double Blind Phase: Placebo (N=8)
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 5 | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 7 | 0 | 0 | 0
Weight increased (Investigations) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Sedation (Nervous system disorders) | 4 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This trial was terminated early due to the withdrawal of post-marketing commitment (PMC) to FDA. The planned interim analysis was not conducted either.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03661983/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT03661983/SAP_001.pdf